CLINICAL TRIAL: NCT04117399
Title: Effect of Inspiratory Muscle Training on Posture in Chronic Obstructive Pulmonary Disease Patients (COPD)
Brief Title: Effect of Inspiratory Muscle Training on Posture in Chronic Obstructive Pulmonary Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Bilel Tounsi, Principal Investigator, Faculty of Medicine, Sousse
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: COPD-POSTURE
Record Dates: First submitted 2019-09-28; First posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; IMT; CoP ML; CoP AP; Posture
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT group (Experimental): Inspiratory muscle training + aerobic exercice
  Interventions: Other: Pulmonary rehabilitation
- Control group (Active Comparator): aerobic exercice
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — The experimental group receives inspiratory muscle training and aerobic exercise. The Active Comparator group received only aerobic exercise group received only aerobic exercise.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a respiratory disease that results in progressive airflow limitation and respiratory distress. Physiopathological features of COPD suggest that people who suffer from this disease have many risk factors for falls that have been identified in older individuals. Risk of falls is multi-factorial and impaired balance has been shown to contribute.

The investigators aimed to demonstrate that, IMT performed during a PRP may improve Postural control in COPD patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease COPD is a preventable and treatable disease. According to the WHO, COPD would be the third leading cause of death by 2030. This disease is characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and associated with an abnormal inflammatory response of the lung to noxious particles or gases. However, emerging data showed that COPD patients demonstrate important deficits in balance and control which associated to a high risk of fall.

Individuals with COPD, especially those with inspiratory muscle weakness, increased their reliance on ankle muscle proprioceptive signals and decreased their reliance on back muscle proprioceptive signals during balance control, resulting in a decreased postural stability compared to healthy controls. These proprioceptive changes may be due to an impaired postural contribution of the inspiratory muscles to trunk stability.

Inspiratory muscle training (IMT) has been shown to be an effective modality for COPD patients for improving the maximal inspiratory muscle strength, the dyspnea and health-related quality of life. However, the effect of inspiratory muscle training on postural control is not studying. The purpose of this study is to evaluate the effect of the inspiratory muscles training on posture in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Were COPD diagnosed by pulmonary function testing
* Clinically stable
* Abscence of other obstructive diseases
* Signed written consert

Exclusion Criteria:

* Were previous pneumonectomy or lobectomy in the past 6 months
* Spontaneous risk of pneumothorax or rib fracture
* Incapacity to follow a standard rehabilitation programme (locomotor deficits, acute cardiac failure and acute exacerbation of COPD at the beginning of the programme)
* Lower limb injury
* Neurological injury or disease
* The absence of written informed consent

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-11-15 (Estimated)

PRIMARY OUTCOMES:
Balance outcomes | Basline, After 2 months
  Balance were measured by stabilometry to evaluate postural control in COPD patients. Two principals variabels were evaluated: the center of pressure in the mediolateral direction (CoP ML) ; the center of presure in anteroposterior direction (CoP AP).

CONTACTS AND LOCATIONS:
Locations (1):
- Bilel TOUNSI, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith MD, Chang AT, Seale HE, Walsh JR, Hodges PW. Balance is impaired in people with chronic obstructive pulmonary disease. Gait Posture. 2010 Apr;31(4):456-60. doi: 10.1016/j.gaitpost.2010.01.022. Epub 2010 Mar 4. PMID 20206529
- [Background] Janssens L, Brumagne S, McConnell AK, Claeys K, Pijnenburg M, Burtin C, Janssens W, Decramer M, Troosters T. Proprioceptive changes impair balance control in individuals with chronic obstructive pulmonary disease. PLoS One. 2013;8(3):e57949. doi: 10.1371/journal.pone.0057949. Epub 2013 Mar 1. PMID 23469255